CLINICAL TRIAL: NCT00907777
Title: Vaccination With the Pneumococcal Vaccine GSK 1024850A or Prevenar™ at Approximately 4 Years of Age in Children Primed With 3 Doses of GSK 1024850A Vaccine or Prevenar™ and Boosted With 23-valent Pneumococcal Plain Polysaccharide Vaccine
Brief Title: Vaccination With GSK 1024850A in Children Primed With GSK 1024850A & Boosted With Pneumovax 23™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 112807; 2008-007605-37 (EudraCT Number)
Record Dates: First submitted 2009-05-21; First posted 2009-05-25 (Estimated); Results first posted 2017-01-06 (Estimated); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Infections, Streptococcal; Streptococcus Pneumoniae
Keywords: Haemophilus influenzae; Streptococcus pneumoniae; safety; Pneumococcal conjugate vaccine; immunogenicity
MeSH Terms: conditions — Streptococcal Infections; Haemophilus Infections

ARMS (2):
- Pn Group (Experimental): Subjects receiving GSK 1024850A vaccine.
  Interventions: Biological: Pneumococcal conjugate vaccine GSK 1024850A
- Prev Group (Active Comparator): Subjects receiving Prevenar™ vaccine.
  Interventions: Biological: Pneumococcal conjugate vaccine Prevenar™ (Wyeth Lederle's)

INTERVENTIONS:
Biological: Pneumococcal conjugate vaccine GSK 1024850A — One dose of vaccine will be injected intramuscularly into the deltoid.
  Arms: Pn Group
Biological: Pneumococcal conjugate vaccine Prevenar™ (Wyeth Lederle's) — One dose of vaccine will be injected intramuscularly into the deltoid.
  Arms: Prev Group

SUMMARY:
The aim of this study is to assess the immune response, safety and reactogenicity following administration of an additional dose of a pneumococcal conjugate vaccine at approximately 4 years of age in children previously vaccinated with 3 primary doses of GSK 1024850A or Prevenar™ vaccine within the first 6 months of life and a booster dose of plain polysaccharide pneumococcal (Pneumovax 23™) vaccine at 11-14 months of age.

Antibody persistence will also be assessed at approximately 4 years of age in children previously vaccinated with 3 doses of either GSK 1024850A or Prevenar™ vaccine followed by a booster dose of Pneumovax 23™.

This protocol posting deals with objectives & outcome measures of the extension phase at year 4. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT 00307541). The objectives & outcome measures of the booster phase are presented in a separate protocol posting (NCT 00333450).

ELIGIBILITY:
Inclusion Criteria:

* Male or female between, and including, 46-50 months of age at the time of vaccination.
* Subjects for whom the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.
* Subjects who previously participated in study NCT00333450 in centres with more than 2 subjects and received a booster dose of Pneumovax 23™.
* Written informed consent obtained from both parents/guardians of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the vaccination, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the vaccination.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting one month before study vaccination and during the entire study period.
* Administration of any pneumococcal vaccine since the end of study NCT00333450.
* Administration of immunoglobulins and/or any blood products less than 3 months prior to the vaccination or planned use during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical
* History of any neurologic disorders or seizures
* Anaphylactic reaction following previous administration of the vaccine or history of reactions or allergic disease likely to be exacerbated by any component of the vaccine.
* History of hypotonic-hyporesponsive episode after any previous vaccination.
* Major congenital defects or serious chronic illness.
* History of invasive pneumococcal diseases.
* Acute disease at the time of vaccination
* Rectal temperature >= 38.0°C or oral/axillary/tympanic temperature >= 37.5°C. A temperature greater than or equal to these cut-offs warrants deferral of the vaccination pending recovery of the subject.

Ages: 46 Months to 50 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2009-06-23 (Actual); Primary Completion 2009-10-05 (Actual); Study Completion 2009-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- Germany (14):
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Nördlingen, Bavaria
  - GSK Investigational Site, Bad Oeynhausen, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Heiligenhaus, North Rhine-Westphalia
  - GSK Investigational Site, Mönchengladbach, North Rhine-Westphalia
  - GSK Investigational Site, Willich, North Rhine-Westphalia
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Bad Lobenstein, Thuringia
  - GSK Investigational Site, Neuhaus am Rennweg, Thuringia
  - GSK Investigational Site, Weimar, Thuringia
  - GSK Investigational Site, Berlin

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=472

REFERENCES:
- [Background] Knuf M, Pankow-Culot H, Grunert D, Rapp M, Panzer F, Kollges R, Fanic A, Habib A, Borys D, Dieussaert I, Schuerman L. Induction of immunologic memory following primary vaccination with the 10-valent pneumococcal nontypeable Haemophilus influenzae protein D conjugate vaccine in infants. Pediatr Infect Dis J. 2012 Jan;31(1):e31-6. doi: 10.1097/INF.0b013e3182323ac2. PMID 21909049
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 112807 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112807 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112807 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112807 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112807 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112807 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Prevnar Group: Subjects who were previously vaccinated with three primary doses of Prevnar™ vaccine in study 2005-003299-40 [10PN-PD-DIT-003 (105554)] and a booster dose of Pneumovax 23™ vaccine in study 2006-000560-93 [10PN-PD-DIT-008 BST: 003 (106623)], received one additional dose of Prevnar™ vaccine, administered intramuscularly in the deltoid, at approximately 4 years of age.
- GSK 1024850A Group: Subjects who were previously vaccinated with three primary doses of GSK 1024850A vaccine in study 2005-003299-40 [10PN-PD-DIT-003 (105554)] and a booster dose of Pneumovax 23™ vaccine in study 2006-000560-93 [10PN-PD-DIT-008 BST: 003 (106623)], received one additional dose of GSK 1024850A vaccine, administered intramuscularly in the deltoid, at approximately 4 years of age.
Period: Overall Study
Arm/Group | Prevnar Group | GSK 1024850A Group
Started | 25 | 27
Completed | 25 | 26
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prevnar Group | GSK 1024850A Group | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Continuous [Mean (Standard Deviation); unit: Months] | 46.6 (0.91) | 46.7 (0.72) | 46.65 (0.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 17 | 26
  Male | 16 | 10 | 26

OUTCOME MEASURES:

1. Primary Outcome: Vaccine Pneumococcal Serotype Antibody Concentrations
Description: The anti-pneumococcal antibody concentration cut-off value assessed was greater than or equal to ≥ 0.05 microgram per milliliter (μg/mL). The vaccine pneumococcal serotypes assessed include 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F, and 23F.
Time Frame: Before (PRE) and one month after (POST) the additional dose
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity endpoint measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Prevnar Group | GSK 1024850A Group
Number analyzed (Participants) | 24 | 26
μg/mL
  ANTI-1 PRE: number analyzed (Participants) | 21 | 24
  ANTI-1 PRE | 0.14 [0.09 to 0.23] | 0.38 [0.25 to 0.56]
  ANTI-1 POST | 0.16 [0.1 to 0.25] | 1.35 [1.05 to 1.73]
  ANTI-4 PRE: number analyzed (Participants) | 21 | 24
  ANTI-4 PRE | 0.27 [0.15 to 0.5] | 0.12 [0.08 to 0.19]
  ANTI-4 POST | 4.3 [3.38 to 5.48] | 6.76 [4.91 to 9.3]
  ANTI-5 PRE: number analyzed (Participants) | 21 | 24
  ANTI-5 PRE | 0.11 [0.08 to 0.16] | 0.5 [0.34 to 0.75]
  ANTI-5 POST | 0.15 [0.1 to 0.22] | 1.78 [1.34 to 2.37]
  ANTI-6B PRE: number analyzed (Participants) | 21 | 23
  ANTI-6B PRE | 0.65 [0.38 to 1.12] | 0.48 [0.26 to 0.88]
  ANTI-6B POST | 7.46 [4.61 to 12.08] | 1.68 [1.1 to 2.56]
  ANTI-7F PRE: number analyzed (Participants) | 21 | 24
  ANTI-7F PRE | 0.18 [0.1 to 0.32] | 0.39 [0.26 to 0.59]
  ANTI-7F POST | 0.19 [0.11 to 0.32] | 2.53 [1.83 to 3.51]
  ANTI-9V PRE: number analyzed (Participants) | 21 | 24
  ANTI-9V PRE | 0.48 [0.27 to 0.86] | 0.44 [0.29 to 0.65]
  ANTI-9V POST | 6.88 [4.98 to 9.51] | 2.13 [1.54 to 2.94]
  ANTI-14 PRE: number analyzed (Participants) | 21 | 24
  ANTI-14 PRE | 1.5 [0.82 to 2.74] | 1.98 [1.14 to 3.42]
  ANTI-14 POST | 25.82 [14.65 to 45.5] | 9.71 [5.61 to 16.82]
  ANTI-18C PRE: number analyzed (Participants) | 21 | 24
  ANTI-18C PRE | 0.34 [0.2 to 0.58] | 0.48 [0.26 to 0.9]
  ANTI-18C POST | 4.23 [2.94 to 6.08] | 6.4 [4.61 to 8.87]
  ANTI-19F PRE: number analyzed (Participants) | 21 | 23
  ANTI-19F PRE | 2.02 [1.29 to 3.16] | 2.37 [1.41 to 3.98]
  ANTI-19F POST | 5.68 [3.82 to 8.45] | 15.61 [11.51 to 21.18]
  ANTI-23F PRE: number analyzed (Participants) | 21 | 24
  ANTI-23F PRE | 0.33 [0.2 to 0.53] | 0.23 [0.12 to 0.43]
  ANTI-23F POST | 5.82 [3.77 to 8.97] | 1.27 [0.9 to 1.8]

2. Secondary Outcome: Opsonophagocytic Activity Against Vaccine Pneumococcal Serotypes
Description: The opsonophagocytic activity cut-off value assessed was greater than or equal to ≥ 8. The vaccine pneumococcal serotypes assessed include 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F, and 23F.
Time Frame: Before (PRE) and one month after (POST) the additional dose
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity endpoint measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Prevnar Group | GSK 1024850A Group
Number analyzed (Participants) | 24 | 26
Titers
  OPSONO-1 PRE: number analyzed (Participants) | 22 | 25
  OPSONO-1 PRE | 4 [4 to 4] | 5.8 [3.6 to 9.4]
  OPSONO-1 POST: number analyzed (Participants) | 24 | 25
  OPSONO-1 POST | 5.5 [3.4 to 9.1] | 49.3 [25.5 to 95.2]
  OPSONO-4 PRE: number analyzed (Participants) | 21 | 23
  OPSONO-4 PRE | 20.7 [6.4 to 67.5] | 12.3 [4.5 to 33.9]
  OPSONO-4 POST | 4814 [3380.8 to 6854.6] | 4380.7 [3020.5 to 6353.4]
  OPSONO-5 PRE: number analyzed (Participants) | 23 | 25
  OPSONO-5 PRE | 4.2 [3.8 to 4.6] | 7.5 [4.5 to 12.5]
  OPSONO-5 POST: number analyzed (Participants) | 24 | 25
  OPSONO-5 POST | 4.4 [3.8 to 5.1] | 50.6 [30.8 to 83]
  OPSONO-6B PRE: number analyzed (Participants) | 22 | 24
  OPSONO-6B PRE | 188.2 [55.5 to 638] | 66.3 [19.7 to 222.7]
  OPSONO-6B POST | 6734.3 [3873.2 to 11708.7] | 1424.5 [775 to 2618.4]
  OPSONO-7F PRE: number analyzed (Participants) | 22 | 24
  OPSONO-7F PRE | 1202.9 [809 to 1788.8] | 1498.9 [1097.8 to 2046.6]
  OPSONO-7F POST | 1304.2 [880.7 to 1931.4] | 4657.1 [3321.2 to 6530.3]
  OPSONO-9V PRE: number analyzed (Participants) | 22 | 23
  OPSONO-9V PRE | 612.9 [458.6 to 819.3] | 442 [224.5 to 870.3]
  OPSONO-9V POST: number analyzed (Participants) | 23 | 26
  OPSONO-9V POST | 5829.4 [3909.1 to 8693.2] | 2843.5 [2016 to 4010.6]
  OPSONO-14 PRE: number analyzed (Participants) | 21 | 25
  OPSONO-14 PRE | 149.7 [65.2 to 343.5] | 330 [186.5 to 584]
  OPSONO-14 POST | 5400.8 [3491.3 to 8354.8] | 2812.4 [1734.3 to 4560.7]
  OPSONO-18C PRE: number analyzed (Participants) | 21 | 24
  OPSONO-18C PRE | 16.1 [5.3 to 49.2] | 23.7 [7.5 to 74.2]
  OPSONO-18C POST: number analyzed (Participants) | 24 | 25
  OPSONO-18C POST | 1615.2 [782 to 3336.1] | 2806.6 [1408.8 to 5591.2]
  OPSONO-19F PRE: number analyzed (Participants) | 22 | 25
  OPSONO-19F PRE | 26.1 [14.8 to 46.1] | 35.8 [18.6 to 68.8]
  OPSONO-19F POST: number analyzed (Participants) | 24 | 25
  OPSONO-19F POST | 241.6 [133.6 to 436.7] | 837.3 [559.5 to 1253.2]
  OPSONO-23F PRE: number analyzed (Participants) | 21 | 25
  OPSONO-23F PRE | 1430.2 [542.5 to 3770.6] | 1383.2 [630.2 to 3036]
  OPSONO-23F POST | 23977.2 [14185.3 to 40528.2] | 4865.1 [3977 to 5951.4]

3. Secondary Outcome: Cross-reactive Pneumococcal Serotype Antibody Concentrations
Description: The anti-pneumococcal antibody concentration cut-off value assessed was greater than or equal to ≥ 0.05 microgram per milliliter (μg/mL). The cross-reactive pneumococcal serotypes assessed include 6A and 19A.
Time Frame: Before (PRE) and one month after (POST) the additional dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Prevnar Group | GSK 1024850A Group
Number analyzed (Participants) | 24 | 26
μg/mL
  ANTI-6A PRE: number analyzed (Participants) | 21 | 24
  ANTI-6A PRE | 0.22 [0.13 to 0.37] | 0.19 [0.12 to 0.32]
  ANTI-6A POST | 1.78 [0.88 to 3.59] | 0.47 [0.29 to 0.75]
  ANTI-19A PRE: number analyzed (Participants) | 21 | 24
  ANTI-19A PRE | 0.39 [0.2 to 0.78] | 0.29 [0.17 to 0.5]
  ANTI-19A POST | 0.8 [0.44 to 1.44] | 1.24 [0.79 to 1.95]

4. Secondary Outcome: Opsonophagocytic Activity Against Cross-reactive Pneumococcal Serotypes
Description: The opsonophagocytic activity cut-off value assessed was greater than or equal to ≥ 8. The cross-reactive pneumococcal serotypes assessed include 6A and 19A.
Time Frame: Before (PRE) and one month after (POST) the additional dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Prevnar Group | GSK 1024850A Group
Number analyzed (Participants) | 24 | 24
Titers
  OPSONO-6A PRE: number analyzed (Participants) | 20 | 22
  OPSONO-6A PRE | 106.9 [44.7 to 255.7] | 117.7 [43.6 to 318.3]
  OPSONO-6A POST: number analyzed (Participants) | 24 | 22
  OPSONO-6A POST | 2320.4 [1180.2 to 4562.5] | 966.2 [634.8 to 1470.6]
  OPSONO-19A PRE: number analyzed (Participants) | 23 | 23
  OPSONO-19A PRE | 10.4 [4.9 to 22.1] | 19.6 [6.6 to 58.8]
  OPSONO-19A POST | 101.3 [42.7 to 240.7] | 153.9 [67.7 to 349.9]

5. Secondary Outcome: Anti-protein D Antibody Concentrations
Description: The anti-protein D antibody cut-off value (greater than or equal to ≥100 EL.U/mL) was assessed by Enzyme-Linked Immuno Sorbent Assay (ELISA) unit per milliliter (EL.U/mL).
Time Frame: Before (PRE) and one month after (POST) the additional dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Prevnar Group | GSK 1024850A Group
Number analyzed (Participants) | 24 | 26
EL.U/mL
  ANTI-PD PRE: number analyzed (Participants) | 21 | 23
  ANTI-PD PRE | 104.1 [76.8 to 140.9] | 173.1 [113.5 to 263.9]
  ANTI-PD POST | 85.9 [64.1 to 115] | 1135.6 [709 to 1819]

6. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness, and swelling. Grade 3 pain was defined as crying when limb was moved/spontaneously painful. Grade 3 swelling/redness was defined as swelling/redness larger (>) 30 millimeters (mm). "Any" is defined as incidence of the specified symptom regardless of intensity.
Time Frame: During the 8-day (Days 0-7) post-additional dose
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with the additional vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Prevnar Group | GSK 1024850A Group
Number analyzed (Participants) | 25 | 26
Participants
  Any Pain | 11 | 16
  Grade 3 Pain | 0 | 2
  Any Redness | 13 | 14
  Grade 3 Redness | 7 | 3
  Any Swelling | 7 | 9
  Grade 3 Swelling | 4 | 1

7. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms assessed include drowsiness, fever (defined as rectal temperature ≥ 38.0°C), irritability, and loss of appetite. Grade 3 drowsiness was defined as drowsiness which prevented normal everyday activities. Grade 3 fever was defined as fever (rectal temperature) above (>) 40.0 degree Celsius (°C). Grade 3 irritability was defined as crying that could not be comforted/preventing normal everyday activities. Grade 3 loss of appetite was defined as the subject not eating at all. "Any" is defined as incidence of the specified symptom regardless of intensity or relationship to study vaccination.
Time Frame: During the 8-day (Days 0-7) post-additional dose
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Prevnar Group | GSK 1024850A Group
Number analyzed (Participants) | 25 | 26
Participants
  Any Drowsiness | 4 | 12
  Grade 3 Drowsiness | 0 | 1
  Related Drowsiness | 0 | 8
  Any Fever | 1 | 8
  Grade 3 Fever | 0 | 0
  Related Fever | 0 | 6
  Any Irritability | 5 | 9
  Grade 3 Irritability | 0 | 1
  Related Irritability | 2 | 7
  Any Loss of appetite | 3 | 12
  Grade 3 Loss of appetite | 0 | 2
  Related Loss of appetite | 1 | 7

8. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. "Any" is defined an incidence of an unsolicited AE regardless of intensity or relationship to study vaccination.
Time Frame: Within 31 days (Day 0-30) post-additional vaccination
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Prevnar Group | GSK 1024850A Group
Number analyzed (Participants) | 25 | 27
Participants | 8 | 6

9. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: An SAE is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or may evolve into one of the outcomes listed above.
Time Frame: Throughout the entire study period (approximately 1 month per subject)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Prevnar Group | GSK 1024850A Group
Number analyzed (Participants) | 25 | 27
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: SAEs: during the entire study period (approximately 1 month per subject); Solicited local and general symptoms: within 8 days after the additional vaccination; Unsolicited symptoms: within 31 days after the additional vaccination.
Arm/Group | Prevnar Group | GSK 1024850A Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 17/25 | 20/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Prevnar Group (N=25) | GSK 1024850A Group (N=27)
Pain (General disorders) | 11 | 16/26
Redness (General disorders) | 13 | 14/26
Swelling (General disorders) | 7 | 9/26
Drowsiness (General disorders) | 4 | 12/26
Fever (>38.0°C) (General disorders) | 1 | 8/26
Irritability (General disorders) | 5 | 9/26
Loss of appetite (General disorders) | 3 | 12/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.